CLINICAL TRIAL: NCT05801445
Title: Increasing Movement and Exercise in Geriatric Patients Through Large-Scaled Creative Occupation Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jason Eugene Vice, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300010109
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Physical Fitness in Older Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupational Arm (Experimental)
  Interventions: Behavioral: Occupation-based activity
- Traditional Exercise Arm (Active Comparator)
  Interventions: Behavioral: Body-Weight Exercise

INTERVENTIONS:
Behavioral: Occupation-based activity — Painting large-scale canvas
  Arms: Occupational Arm
Behavioral: Body-Weight Exercise — Body-weight exercises designed for older adults
  Arms: Traditional Exercise Arm

SUMMARY:
The goal of this clinical trial is to compare two different types of activities in improving physical fitness in older adults. The main question it aims to answer is whether a person completing a large-scaled art project has similar physical improvements as a person completing a more traditional exercise program.

Participants will be asked to either stand for up to an hour while completing a painting across a large canvas or stand for up to an hour while doing body weight exercises. Researchers will compare the painting group to the exercise group to see if physical improvements are the same or different.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether large-scaled creative occupations, such as painting large paintings, would be equally, if not more beneficial than traditional exercise for older adults. Painting on large mural-sized paintings will simulate the participation of endurance heavy, physically demanding tasks. This is because to complete the task, participants will be required to reach to cover the canvas, stand for extended periods of time, and perform repetitive movements. It is hypothesized that this activity will increase active range of motion, strength, endurance, balance, as well as motivation to participate in physical activity by providing a more enjoyable, alternative form of exercise.

ELIGIBILITY:
Exclusion Criteria:

* Individuals unable to stand with minimal support

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Upper extremity active range of motion | 10 weeks
  Degrees goniometry
Upper and lower extremity strength | 10 weeks
  Manual muscle test
Standing balance | 10 weeks
  Functional reach test

SECONDARY OUTCOMES:
Self-motivation | 10 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Crowne Health Services, Citronelle, Alabama, United States

IPD SHARING:
Plan to Share IPD: No